CLINICAL TRIAL: NCT01244542
Title: Pain and Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4706
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Pain; Schizophrenia
Keywords: Schizophrenia; DSM IV criteria; Pain insensitivity; Painful perception; Opioid receptors
MeSH Terms: conditions — Pain; Schizophrenia; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with schizophrenia (Experimental)
  Interventions: Other: unpleasant stimuli
- Healthy controls (Active Comparator): controls matched with patients on age, sex and education level
  Interventions: Other: unpleasant stimuli

INTERVENTIONS:
Other: unpleasant stimuli

SUMMARY:
The aim of the investigators project is to explore the mechanisms of pain insensitivity in patients with schizophrenia, in order to prevent its invalidating consequences. The investigators will couple methods of experimental psychology with EEG and blood samplings, in order to distinguish the role of non-painful perception, attention, aversive effects, and pain expression, and the investigators will explore an original neurobiological hypothesis regarding the activation of opioid receptors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia (criteria DSM IV) or healthy controls matched with patients on age, sex and education level
* 18-55 years old

Exclusion Criteria:

* Past history affecting CNS
* Intake of psychotropic drugs, except for patients
* Metabolic disorder affecting sensory processing (diabetes)
* Intake of benzodiazepines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Unpleasant stimuli | during experimental session
  acute electrical stimulation
Unpleasant stimuli | during experimental session
  emotional pictures

CONTACTS AND LOCATIONS:
Overall Officials: Anne Giersch, MD, Study Director — University Hospital, Strasbourg, France
Locations (5):
- France (5):
  - Service de Psychiatrie Adulte2, Place Saint-Jacques - ZA 481, Centre Hospitalier Saint-Jacques, Besançon
  - Service de Psychiatrie Adulte, Secteur G11, Centre Hospitalier de Erstein, 13 route de Krafft, Erstein
  - Centre d'évaluation et de traitement de la douleur, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre d'Investigation Clinique - Hôpitaux Universitares de Strasbourg, Strasbourg
  - Service de Psychiatrie - Hôpitaux Universitaires de Strasbourg, Strasbourg